CLINICAL TRIAL: NCT06038838
Title: Evaluation of Safety and Feasibility of the Tioga TMVR System for Treatment of Mitral Regurgitation
Brief Title: Feasibility Study of the Tioga TMVR System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tioga Cardiovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-03218
Record Dates: First submitted 2023-08-30; First posted 2023-09-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Patients with Symptomatic MR (MR>=3+) (Experimental): Subjects treated with the Tioga TMVR System
  Interventions: Device: Tioga TMVR System

INTERVENTIONS:
Device: Tioga TMVR System — A bioprosthetic mitral valve, as part of the Tioga TMVR System, is implanted percutaneously in a patient with MR via transfemoral-transseptal access.

SUMMARY:
The study is aimed to assess the safety and feasibility of the Tioga TMVR System in treating patients with symptomatic MR (MR>=3+)

DETAILED DESCRIPTION:
The Tioga TMVR Feasibility Study is a prospective, single-arm, multi-center study with a planned enrollment of up to 30 patients. The Tioga TMVR System is designed to percutaneously replace a patient's diseased native mitral valve with a bioprosthetic valve. The investigational device is intended for transseptal replacement of the mitral valve in patients with symptomatic MR (MR>=3+).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Symptomatic, moderate to severe (3+) or severe (4+) MR
* NYHA Functional Classification ≥ II
* Heart team concurs that the subject is non-ideal for surgical intervention or other available treatment options (e.g., TEER)
* The subject or the subject's legal representative has been informed of the nature of the study, has agreed to return for post-procedure follow-up visits, and has provided informed consent

Exclusion Criteria:

* LVEF < 30%
* LVEDD > 70 mm
* Anatomic features (e.g., annular dimensions, neo-LVOT area, transfemoral and transseptal access, MAC) unsuitable for the Tioga TMVR System
* Severe aortic valve stenosis or regurgitation
* Severe right ventricular dysfunction or severe tricuspid valve disease
* Evidence of intracardiac thrombus, vegetation, or mass
* Prior mitral valve intervention
* Prior prosthetic heart valve in any position
* Any percutaneous coronary, carotid, or other endovascular intervention within 30 days prior to enrollment
* Any carotid surgery within 30 days prior to enrollment
* Any open cardiac or vascular surgery (other than carotid surgery) within 90 days prior to enrolment
* Myocardial infarction within 30 days prior to enrollment
* Cardiac resynchronization therapy (CRT) device implanted within 30 days of enrollment
* History of endocarditis within 6 months prior to enrollment or evidence of active systemic infection or sepsis.
* Planned cardiovascular procedure within 30 days of enrolment
* Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 30 days of enrollment
* Active peptic ulcer or active GI bleeding within 90 days of enrollment
* Cardiogenic shock or hemodynamic instability requiring inotropic support or mechanical heart assistance
* Pulmonary arterial hypertension with fixed PASP > 70mmHg or PVR > 5WU that cannot be reduced to less than 5WU with vasodilator therapy
* Severe chronic obstructive pulmonary Disease (COPD) or airways disease requiring continuous home oxygen
* Renal insufficiency (eGFR <20 mL/min) or ESRD on dialysis
* Life expectancy < 12 months
* Subject is on the waiting list for a transplant or has had a prior heart transplant
* Child class C cirrhosis
* Blood dycrasias as defined by acute anemia with Hb < 9, platelets < 75K, WBC < 0.5
* Female subjects who is breast feeding or pregnant or planning to become pregnant within the study period.
* Known hypersensitivity or contraindication to procedural, post procedural medication (e.g., contrast solution) or hypersensitivity to nickel or titanium
* Inability to tolerate anticoagulation or antiplatelet therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | From index procedure (Day 0) to 30 days post-procedure
  Number of subjects with all-cause mortality, cardiovascular-related hospitalizations, disabling stroke, and/or mitral valve reintervention or reoperation through 30 days post-procedure
Primary Performance Endpoint | At completion of index procedure (Day 0)
  Number of subjects achieving MVARC technical success - all of the following must be present at exit of catheterization lab:
  * Absence of procedural mortality
  * Successful access, delivery, and retrieval of the device delivery system
  * Successful deployment and correct positioning of the first intended device
  * Freedom from emergency surgery or reintervention related to the device or access procedure

CONTACTS AND LOCATIONS:
Locations (5):
- Incor - Instituto do Coração do Hospital das Clínicas da FMUSP, São Paulo, Brazil
- Georgia (2):
  - Helsicore Hospital (Israeli Georgeian Medical Research Clinic Healthycore), Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
- Vilnius Univ. Hospital, Vilnius, Lithuania
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: Undecided